CLINICAL TRIAL: NCT06411873
Title: The Effect of High Protein Enteral Nutrition on Critically Ill Postoperative Children: A Study of Nitrogen Balance and Intestinal Fatty Acid Binding Protein
Brief Title: The Effect of High Protein Enteral Nutrition on Critically Ill Postoperative Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Irene Yuniar, Sp.A(K), Lecturer of Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24779
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Enteral Nutrition; Postoperative; Critically Ill Children
Keywords: Proteins; Enteral; Critically ill children; Postoperative
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This trial is an interventional study with two arms. Participants will be randomised to high enteral protein or standard enteral protein. For both trial arms, participants will be provided with enteral nutrition (EN) as per standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were recruited through consecutive sampling until the required number of participants was reached. They were then randomly assigned into study groups using block randomization. The randomization process was conducted online via https://www.sealedenvelope.com/, overseen by the methodology team. Results were stored securely, inaccessible to researchers. Allocation concealment was ensured with sequentially numbered sealed opaque envelopes, indicating standard or high-protein enteral nutrition. These were handed to a designated nutritionist coordinator, independent of the research team, responsible for storage, preparation, and distribution. Research assistants informed the coordinator of subjects, who then prepared the assigned nutrition accordingly. High-protein enteral nutrition resembled standard nutrition to maintain blindness. Researchers, patients, families, nurses, and physicians remained unaware of the nutrition type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The patients included in the control group received the customary protein amount and were fed a standard formula (Pediacomplete, Abbot, Indonesia)
  Interventions: Dietary Supplement: Control Group
- Intervention Group (Experimental): The patients included in the intervention group received the same formula like control group with the addition of modular protein supplement PURO ISOPRO WPI Whey Isolate PLAIN, Puro Pure Nutrition, Sukoharjo, Indonesia (BPOM : MD 862312050010)
  Interventions: Dietary Supplement: Intervention Group

INTERVENTIONS:
Dietary Supplement: Control Group — Composition of formula per 100 mL : energy (100 kcal), protein (3 g), carbohydrate (13.54 g), lipids (3.93 g), protein energy ratio/PER 12%, osmolarity (310 mOsm/L), renal solute load/RSL (27.5 mOsm/100 kcal)
  Arms: Control Group
Dietary Supplement: Intervention Group — Composition of formula per 100 mL : energy (105.5 kcal), protein (4.35 g), carbohydrate (13.54 g), lipids (3.93 g), protein energy ratio/PER 16.5%, osmolarity (333.5 mOsm/L), renal solute load/RSL (27.7 mOsm/100 kcal)
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is o determine the feasibility and efficacy of high enteral protein in critically ill postoperative children. It will also learn about the safety of high enteral protein for critically ill postoperative children. The main questions it aims to answer are:

Does high enteral protein improve nitrogen balance in critically ill postoperative children? Does high enteral protein reduce levels of Intestinal Fatty Acid Binding Protein (I-FABP) in critically ill postoperative children?

Researchers will compare high enteral protein to a standard enteral protein to see if high enteral protein works to improve nitrogen balance and reduces levels of Intestinal Fatty Acid Binding Protein (I-FABP) in critically ill postoperative children.

Participants will:

Take high enteral protein or standard enteral protein for 72 hours The nitrogen balance and I-FABP levels will be assessed both before and after enteral feeding.

Monitoring and reporting of adverse events and serious adverse events will be conducted in accordance with good clinical practice guidelines.

DETAILED DESCRIPTION:
Postoperative care in critically ill children often involves careful attention to nutritional support to optimize recovery and outcomes. Among the various nutritional interventions, high protein enteral nutrition has gained significant attention for its potential benefits in this population. Adequate protein intake is essential for wound healing, immune function, and muscle preservation, all of which are crucial aspects of recovery following surgery in critically ill children.

High protein enteral nutrition offers a targeted approach to meet the increased protein requirements during the postoperative period. By providing a concentrated source of protein directly into the gastrointestinal tract, it bypasses potential barriers associated with oral intake and facilitates nutrient absorption in a controlled manner. Additionally, enteral nutrition is preferred over parenteral nutrition due to its lower risk of complications and potential to maintain gut integrity and function.

Despite its theoretical advantages, the clinical efficacy of high protein enteral nutrition in critically ill postoperative children remains an area of ongoing research. Studies investigating its impact on nitrogen balance, muscle protein synthesis, immune function, and clinical outcomes are essential for guiding nutritional practices in this vulnerable population.

This study aim to evaluate the effect of high protein enteral nutrition on critically ill postoperative children, with a focus on assessing nitrogen balance and intestinal fatty acid binding protein levels. Through comprehensive analysis, potential benefits and challenges associated with this nutritional intervention will be identified, ultimately informing evidence-based nutritional strategies for optimizing postoperative care in critically ill pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill postoperative children (age 1 to 5 years of age)
2. Hemodynamically stable within 48 hours postoperative
3. The patient receives enteral nutrition within 48 hours postoperative
4. The patient can undergo observation and examination for up to 72 hours after enteral nutrition therapy
5. The parents/guardians are willing to participate in the study by signing the informed consent

Exclusion Criteria:

1. Patients with absolute contraindications (paralytic/mechanical ileus, gastrointestinal obstruction, gastrointestinal perforation) or relative contraindications (gastrointestinal dysmotility, necrotizing enterocolitis, toxic megacolon, extensive peritonitis, gastrointestinal bleeding, gastrointestinal fistula) to enteral nutrition administration.
2. Patients with a history of cow's milk allergy or using special formula milk.
3. Patients still receiving breast milk (breastfeeding).
4. Patients at high risk of refeeding syndrome according to ASPEN consensus
5. Patients with acute or chronic kidney disorders.
6. Patients with liver disorders.
7. Patients with diabetes mellitus.
8. Patients with inborn errors of metabolism.
9. Patients receiving total parenteral nutrition.
10. Patients requiring continuous life support devices such as continuous renal replacement therapy (CRRT) or extracorporeal membrane oxygenation (ECMO).
11. Nitrogen balance cannot be measured (patients with drainage production >1 ml/kg/hour or bleeding >10% of total blood volume at the time of enteral nutrition initiation).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Nitrogen Balance | Nitrogen balance will be assessed both before and after 72 hours enteral feeding
  The Nitrogen Balance was calculated by subtracting nitrogen losses from the nitrogen intake, including urinary, faecal and miscellaneous losses (dermal, sweat, integumentary) with the following formula:
  Nitrogen Balance (mg/kg) = nitrogen intake (mg/kg) -(total urine nitrogen (mg/kg) + 75 mg/kg) where 75 mg/kg represents faecal and miscellaneous nitrogen losses. The total urinary nitrogen (TUN) excretion was estimated as the urinary urea nitrogen (UUN) concentration (mg/kg) × 1.25 to include nitrogen losses in the form of ammonia, creatinine, uric acid and amino acids. The UUN check from 24 hours urine sample.
I-FABP Levels | I-FABP levels will be assessed both before and after 72 hours enteral feeding
  The blood samples for measuring I-FABP levels (pg/mL) will be securely transported to and processed at Prodia Laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided